CLINICAL TRIAL: NCT00750529
Title: Effects of Galantamine and Donépézil on the Amount and the Quality oh the Sleep in Patients Suffering From Alzheimer Disease.
Brief Title: Alzheimer and Sleep
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Janssen-Cilag Farmaceutica Ltda. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0038
Record Dates: First submitted 2008-09-09; First posted 2008-09-10 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Alzheimer's Disease
Keywords: sleep; Alzheimer; old patients
MeSH Terms: conditions — Alzheimer Disease | interventions — Galantamine; Donepezil

ARMS (1):
- Galantamine (Experimental)
  Interventions: Drug: Galantamine and Donepezil

INTERVENTIONS:
Drug: Galantamine and Donepezil — the analysis of two inhibitors of Ach-E : galantamine and donézepil in over 65 years old patients suffering from Alzheimer's disease (MMSE between 20 and 26) without Alzheimer's medication

SUMMARY:
The aim of the study is the analysis of two inhibitors of Ach-E: galantamine and donépézil in over 65 years' old patients suffering from Alzheimer disease (MMSE between 20 and 26) without Alzheimer's medication.

DETAILED DESCRIPTION:
Feasibility study, open, randomized, controlled, cross-over study in 65 years old patients.

ELIGIBILITY:
Inclusion Criteria:

* 65 and over years old
* Patients suffering from Alzheimer disease
* Patient living with someone at home
* Written consent given

Exclusion Criteria:

* Galantamine or Donepezil hypersensibility
* Patient living alone and in a medicalized structure
* Concomitant medication
* Chronical diseases

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-11; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Comparison of the percentage of paradoxical sleep recorded with polysomonography in 65 years old patients with administration of Galantamine or Donépézil | administration of galantamine or donépézil

SECONDARY OUTCOMES:
Describe the iatrogenic modifications of rhythm and architecture of sleep. describe the iatrogenic modifications of rythm and architecture of sleep | during the iatrogenic modifications

CONTACTS AND LOCATIONS:
Overall Officials: Dubray Claude, Pr, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (2):
- France (2):
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CPC-CIC, Clermont-Ferrand